CLINICAL TRIAL: NCT04791592
Title: Pecto-Intercostal Fascial Block Versus Transversus Thoracic Muscle Plane Block for Acute Post-sternotomy Pain After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study
Brief Title: Pecto-Intercostal Fascial Block vs. Transversus Thoracic Muscle Plane Block in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cengiz KAYA, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PIFB-TTPB19
Record Dates: First submitted 2021-03-09; First posted 2021-03-10 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Pain, Postoperative; Coronary Artery Disease
Keywords: Pain, Postoperative; Surgery, Cardiac; Nerve, Block
MeSH Terms: conditions — Pain, Postoperative; Coronary Artery Disease; Bites and Stings

STUDY DESIGN:
Intervention Model Description: The patients will be randomly classified into two groups.
Who Masked: Participant, Investigator
Masking Description: Patients randomly will be classified into two groups using opaque sealed envelopes. Randomization will be performed using a computer-generated random number list, and a statement indicating the patient's group is placed in a closed envelope numbered according to the result. Each patient will be asked to choose an envelope, and the patients will be assigned to the study according to the group written in the envelope. An anesthesiologist with expertise in regional anesthesia will perform PIF and TTP block to ensure the block's quality and consistency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PIFB (Active Comparator): PIF block (20 ml, 0.25% bupivacaine + 1:400.000 adrenaline) + IV morphine-PCA
  Interventions: Procedure: Single-injection, ultrasound-guided bilateral PIF block.
- Group TTMPB (Active Comparator): TTMP block (20 ml, 0.25% bupivacaine + 1:400.000 adrenaline) + IV morphine-PCA
  Interventions: Procedure: Single-injection, ultrasound-guided bilateral TTMP block.

INTERVENTIONS:
Procedure: Single-injection, ultrasound-guided bilateral PIF block. — PIF block bilaterally (20 ml, 0.25% bupivacaine + 1:400.000 adrenaline). In addition, LA infiltration (10 ml, 0.25% bupivacaine) will be performed by the surgeon around the chest tube in all patients.
  Intraoperative analgesia: At the end of the surgery, all patients will be given 0.05 mg/kg morphine IV.
  Postoperative analgesia: Paracetamol 1 gr IV (every 6 hours) and IV PCA of 0.5 mg/ml morphine (demand dose 20µg/kg; lock out interval 6-10 min.; the 4-hour limit will be 80% of the total calculated dose).
  In cases where rescue analgesia is required (NRS score ≥4) tramadol 100 mg IV will be infused within 30 minutes (max. 300 mg / day).
  For postoperative nausea and vomiting prophylaxis, patients will be routinely administered ondansetron 4 mg IV 20 minutes before extubation in the intensive care unit.
  Arms: Group PIFB
Procedure: Single-injection, ultrasound-guided bilateral TTMP block. — TTMP block bilaterally (20 ml, 0.25% bupivacaine + 1:400.000 adrenaline). In addition, LA infiltration (10 ml, 0.25% bupivacaine) will be performed by the surgeon around the chest tube in all patients.
  Intraoperative analgesia: At the end of the surgery, all patients will be given 0.05 mg/kg morphine IV.
  Postoperative analgesia: Paracetamol 1 gr IV (every 6 hours) and IV PCA of 0.5 mg/ml morphine (demand dose 20µg/kg; lock out interval 6-10 min.; the 4-hour limit will be 80% of the total calculated dose).
  In cases where rescue analgesia is required (NRS score ≥4) tramadol 100 mg IV will be infused within 30 minutes (max. 300 mg / day).
  For postoperative nausea and vomiting prophylaxis, patients will be routinely administered ondansetron 4 mg IV 20 minutes before extubation in the intensive care unit.
  Arms: Group TTMPB

SUMMARY:
In patients undergoing open cardiac surgery, pain control is an essential part of the enhanced recovery process. The current study aimed to evaluate the analgesic efficacies of ultrasound-guided pecto-intercostal fascial block and ultrasound-guided transversus thoracic muscle plane block for open cardiac surgeries. Analgesic efficacy will be assessed on the numeric rating scale (NRS) along with intraoperative and 24 h postoperative opioid consumption.

DETAILED DESCRIPTION:
It has been reported that the TTMP block and PIF block produce effective postoperative analgesia for open cardiac surgeries.

The hypothesis of our study; PIF block reduces pain and analgesic consumption in the acute period (0-24 hours) similar to TTP block in patients undergoing elective cardiac surgery requiring median sternotomy.

Patients will be divided into two groups:

Group PIFB: A bilateral PIF block will be performed intraoperatively (20 ml, %0.25 bupivacaine + 1:400.000 adrenaline). In addition, IV morphine patient-controlled analgesia (PCA) will be applied postoperatively for 24 hours.

Group TTMPB: A bilateral TTMP block will be performed intraoperatively (20 ml, %0.25 bupivacaine + 1:400.000 adrenaline). In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients between the ages of 18-80 who are scheduled for elective cardiac surgery (coronary artery bypass graft surgery with median sternotomy +/- valve replacement or isolated valve surgery)
* BMI <35 kg / m2

Exclusion Criteria:

* Emergent surgeries, redo cases, minimally invasive procedures
* Patients who do not want to participate
* Patients with cognitive dysfunction (patients who are not able to evaluate the verbal numerical pain scale)
* Hypersensitivity or history of allergies to local anesthetics
* Patients with severe major organ dysfunction (such as renal or hepatic insufficiency)
* LVEF <30
* Patients with psychiatric disorders
* Pregnancy or breastfeeding
* Presence of hematological disease
* Patients with alcohol-drug addiction
* Patients who use daily opioids for any reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours after surgery | Postoperative day 1
  Morphine consumption in the first 24 hours will be measured by IV PCA. Patients will be able to request opioids via a PCA device when their NRS score is above 3.

SECONDARY OUTCOMES:
Postoperative pain: NRS score | Postoperative Day 1
  Pain status at rest and while coughing will be assessed by NRS scores at 0, 3, 6, 12, 18, and 24 hours after extubation.In addition, the time until first analgesic requirement will be recorded. The NRS is an 11-point numeric scale which ranges from 0 to 10.
Postoperative nausea and vomiting (PONV) | Postoperative Day 1
  The patients will be verbally evaluated according to a descriptive five-point PONV scale at 0, 3, 6, 12, 18, and 24 hours after extubation. If a score of 3 or more is registered, ondansetron 4 mg IV will be administered and repeated after 8 hours if required.The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once; and 4 = vomiting more than once.
Patient satisfaction | Postoperative Day 1
  Patients' satisfaction with pain management will be evaluated with a 5-point verbal satisfaction scale at the end of 24 hours. The Likert scale is 5 = very satisfied, 4 = satisfied, 3 = unsure, 2 = dissatisfied, 1 = very dissatisfied.
The number of patient required rescue analgesic | Postoperative Day 1
  The number of patient requires rescue analgesic will be recorded at 0, 3, 6, 12, 18, and 24 hours after extubation.
Time to extubation | Postoperative Day 1
  After the operation, the time until the patient is extubated will be recorded.
Length of stay in the ICU | The time from admission to the ICU to the time of discharge to the hospital ward; during the hospital stay, an average of 7 days
  Total duration of stay in ICU will be recorded.
Length of stay in the hospital | Measured in days admitted in the hospital, an average of 7 days
  Their stay in the hospital will be recorded.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients have any complications -directly related to the block or the drug used in the block- will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Karakaya, Study Director — Ondokuz Mayıs University
Locations (1):
- Burhan Dost, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khera T, Murugappan KR, Leibowitz A, Bareli N, Shankar P, Gilleland S, Wilson K, Oren-Grinberg A, Novack V, Venkatachalam S, Rangasamy V, Subramaniam B. Ultrasound-Guided Pecto-Intercostal Fascial Block for Postoperative Pain Management in Cardiac Surgery: A Prospective, Randomized, Placebo-Controlled Trial. J Cardiothorac Vasc Anesth. 2021 Mar;35(3):896-903. doi: 10.1053/j.jvca.2020.07.058. Epub 2020 Jul 24. PMID 32798172
- [Background] Kelava M, Alfirevic A, Bustamante S, Hargrave J, Marciniak D. Regional Anesthesia in Cardiac Surgery: An Overview of Fascial Plane Chest Wall Blocks. Anesth Analg. 2020 Jul;131(1):127-135. doi: 10.1213/ANE.0000000000004682. PMID 32032103
- [Background] Caruso TJ, Lawrence K, Tsui BCH. Regional anesthesia for cardiac surgery. Curr Opin Anaesthesiol. 2019 Oct;32(5):674-682. doi: 10.1097/ACO.0000000000000769. PMID 31356362
- [Background] Smith LM, Barrington MJ; St Vincent's Hospital, Melbourne. Ultrasound-guided blocks for cardiovascular surgery: which block for which patient? Curr Opin Anaesthesiol. 2020 Feb;33(1):64-70. doi: 10.1097/ACO.0000000000000818. PMID 31833864
- [Background] Markham T, Wegner R, Hernandez N, Lee JW, Choi W, Eltzschig HK, Zaki J. Assessment of a multimodal analgesia protocol to allow the implementation of enhanced recovery after cardiac surgery: Retrospective analysis of patient outcomes. J Clin Anesth. 2019 May;54:76-80. doi: 10.1016/j.jclinane.2018.10.035. Epub 2018 Nov 6. PMID 30412813
- [Result] Aydin ME, Ahiskalioglu A, Ates I, Tor IH, Borulu F, Erguney OD, Celik M, Dogan N. Efficacy of Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Postoperative Opioid Consumption After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2996-3003. doi: 10.1053/j.jvca.2020.06.044. Epub 2020 Jun 18. PMID 32665179